CLINICAL TRIAL: NCT04997330
Title: Evaluation of Bilateral HF-rTMS Over DLPFC in add-on to Usual Treatment on Abstinence in Alcohol Use Disorder Patients With Executive Dysfunction After Withdrawal
Brief Title: Evaluation of Bilateral HF-rTMS on Abstinence in Alcohol Use Disorder Patients With Executive Dysfunction
Acronym: STIM-ALC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APHP180582; 2020-A00548-31 (Other: N° IDRCB)
Record Dates: First submitted 2021-07-31; First posted 2021-08-09 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-03

CONDITIONS: Alcohol Withdrawal
Keywords: alcool; rTMS; executive; dysfunction; addiction
MeSH Terms: conditions — Behavior, Addictive | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active rTMS (Experimental): Bilateral high frequency (20Hz) Repetitive Transcranial Magnetic Stimulation (rTMS) over DLPFC
  Interventions: Device: Active rTMS
- Sham rTMS (Placebo Comparator): Sham bilateral high frequency (20Hz) Repetitive Transcranial Magnetic Stimulation (rTMS) over DLPFC
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: Active rTMS — Bilateral high frequency (20Hz) rTMS will be delivered (over dorsolateral prefrontal cortex), at two daily sessions (left side on the morning and right side on the afternoon), 10 consecutive days on working day, 1500 pulses/session, 110% of motor threshold determined, 30 trains, 50 pulses per train and 15s inter train. A session will typically last around 10 minutes. Alcohol cues consisted of a selection of 60 alcohol-related pictures (beverage, drinking-related behaviors, alcohol-related cues) from the Geneva Appetitive alcohol Pictures will be presented during each rTMS session.
  Other Names: Experimental group
  Arms: Active rTMS
Device: Sham rTMS — Sham rTMS will be delivered (over dorsolateral prefrontal cortex) , at two daily sessions (left side on the morning and right side on the afternoon), 10 consecutive working days. A session will typically last around 10 minutes. Alcohol cues consisted of a selection of 60 alcohol-related pictures (beverage, drinking-related behaviors, alcohol-related cues) from the Geneva Appetitive alcohol Pictures will be presented during each rTMS session.
  Other Names: Control group
  Arms: Sham rTMS

SUMMARY:
High frequency repetitive transcranial magnetic stimulation (HF-rTMS) over dorsolateral prefrontal cortex (DLPFC) could correct defective executive functions over the hyperactive reward circuit through the meso-fronto-limbic connections. The restored cortical inhibitory control over compulsive alcohol use, could improve abstinence after withdrawal. The goal of this study is to evaluate the efficacy of HF-rTMS over DLPFC in AUD patients with executive dysfunction after withdrawal.

DETAILED DESCRIPTION:
PARTICIPANTS:

Participants with AUD (moderate to mild according to Alcohol Dependance Scale) with executive dysfunctions will be randomized.

DESIGN:

This study is a multicenter pilot double blind randomized controlled trial. After at least seven days of alcohol residential detoxification, executive dysfunctions's participants will be tested. 64 of them with executive dysfunctions will be randomized either in the active rTMS group or in the sham rTMS group. TMS will be performed during hospitalisation over 10 days. rTMS are proposed as an add on to the usual treatment.

INTERVENTION:

20 rTMS (twice a day) will be performed 10 consecutive working days. The target of the rTMS will be the DLPFC (left side in the morning, right side in the afternoon). During each rTMS sessions (active and sham), alcohol related pictures from the Geneva Appetitive alcohol Pictures will be presented.In the active arm, rTMS will be performed with high frequency (20hz, 1500 pulses per session, 110% of motor threshold).In the control group, sham rTMS will be performed.

Participants will be follow up to three months after the end of rTMS treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-75 years
* Alcohol use disorder according to DSM 5, moderate to mild according to ADS
* Residential stay for alcohol detoxofication

Exclusion Criteria:

* Cognitive deficits defined by MoCA <25 (Montreal Cognitive Assessment) performed at least 7days after alcohol detoxification and after at least 12 hours after benzodiazepine cessation
* History of cerebral stroke
* DSM-5 substance use disorders other than nicotine and alcohol
* Contraindication for rTMS :

  * Pregnancy
  * History of epilepsy or seizure
  * Cochlear implants
  * Cardiac pacemaker or intracardiac lines, or metal in the body
* Clinical history of complicated withdrawal symptoms
* History of severe head trauma followed by loss of consciousness
* Actual major depressive episode, schizophrenia according to the MINI (Mini International Neuropsychiatric Interview)
* Breastfeeding women
* Actual or history of organic failure including cirrhosis
* Absence of health insurance; or patient with AME
* Legal protection (curatorship or tutorship)
* Deprive of freedom or security measure
* No adequate mastering of the French language or no ability to consent
* Major socio-economic problem: homelessness
* No written informed consent
* Participation in another interventional study

Secondary inclusion criteria (before randomization):

- Abnormal executive function defined as at least 3 impaired measurements among 19 measurements of 7 tests (Stroop test, Wisconsin test; Trail making test, verbal fluency, 6 elements, Brixton test, Dual task Baddeley test) from the Greffex battery. Each measure will be considered as impaired if it is below 1.65 SD. The procedure and the measurement are standardized. The neuropsychological evaluation will be performed at least seven days after alcohol detoxification and after at least 12 hours after benzodiazepine cessation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with continuous complete alcohol abstinence | 1 month after the end of rTMS sessions
  Percentage of patients with continuous complete abstinence up to one month after the end of the rTMS treatment.
  The abstinence will be assessed using the Alcohol-Time Line Follow Back tool (TLFB). The Alcohol TLFB is a descriptive questionnaire, using a calendar, participants will retrospectively record at M1 the number of days they drank over the 30 days following the end of the rTMS treatment. Continuous complete abstinence will be defined as no day with alcohol consumption over the 30 days.

SECONDARY OUTCOMES:
Percentage of participants with alcohol continuous complete abstinence | 3 months after the end of rTMS sessions
  Percentage of patients with continuous complete abstinence up to 3 months after the end of the rTMS treatment.
  The abstinence will be assessed using the Alcohol-TLFB at M1, M2, M3. Continuous complete abstinence will be defined as no day with alcohol consumption over the 90 days.
Number of cumulative abstinence days | 1 month after the end of rTMS sessions
  Alcohol consumption measured by the number of cumulative abstinence days up to 1 month after the end of the rTMS treatment. The number of cumulative abstinence days will be assessed using (TLFB) at M1 and will be calculated by summing the total number of days when no alcohol was consumed over the 30 days.
Number of cumulative abstinence days | 3 months after the end of rTMS sessions
  Alcohol consumption measured by the number of cumulative abstinence days up to 3 months after the end of the rTMS treatment. The number of cumulative abstinence days will be assessed using (TLFB) at M1, M2, M3 and will be calculated by summing the total number of days when no alcohol was consumed over the 90 days.
Time until the first heavy drinking days (HDD) | 3 months after the end of rTMS sessions
  Time until the first heavy drinking days (HDD) up to 3 months. The time, in days, until the first HDD will be assessed using (TLFB) at M1, M2, M3. HDD will be defined as more than 50 (men) or 40 (women) g/day.
Number of heavy drinking days (HDD) | 1 month after the end of rTMS sessions
  Number of heavy drinking days (HDD) up to 1 month. Number of heavy drinking days HDD will be assessed using (TLFB) at M1 and will be calculated by summing the total number of days with HDD over the 30 days. HDD will be defined as more than 50 (men) or 40 (women) g/day.
Number of heavy drinking days (HDD) | 3 month after the end of rTMS sessions
  Number of heavy drinking days (HDD) up to 3 months. Number of heavy drinking days HDD will be assessed using (TLFB) at M1, M2, M3 and will be calculated by summing the total number of days with HDD over the 90 days.. HDD will be defined as more than 50 (men) or 40 (women) g/day.
Time to relapse | 3 months after the end of rTMS sessions
  The time to relapse, in days, will be assessed using (TLFB) at M1, M2, M3. Relapse will be defined as a day with a consumption equal or higher than 50% of initial intake.
Alcohol dependence severity assessed by the Alcohol Dependence Scale (ADS) | 1 month after the end of rTMS sessions
  Alcohol dependence severity will be evaluated with the Alcohol Dependence Scale (ADS). The ADS is a self-administrated 25-items questionnaire (requiring 5 minutes) assessing alcohol withdrawal symptoms, impaired control over drinking, awareness of compulsive drink, increased tolerance and salience of drink-seeking behavior. ADS is initially used to assess a past 12-month period, its instructions can be modified for different time-frame. The ADS will be assessed on previous 4 weeks. This scale is scored out of 47, higher scores are considered worse.
Alcohol dependence severity assessed by the Alcohol Dependence Scale (ADS) | 3 months after the end of rTMS sessions
  Alcohol dependence severity will be evaluated with the Alcohol Dependence Scale (ADS). The ADS is a self-administrated 25-items questionnaire (requiring 5 minutes) assessing alcohol withdrawal symptoms, impaired control over drinking, awareness of compulsive drink, increased tolerance and salience of drink-seeking behavior. ADS is initially used to assess a past 12-month period, its instructions can be modified for different time-frame. The ADS will be assessed on previous 4 weeks. This scale is scored out of 47, higher scores are considered worse.
Alcohol cue induced craving using the Cue induced Obsessive Compulsive Drinking Scale (OCDS) | At the last day of rTMS sessions
  Evaluated by Cue induced Obsessive Compulsive Drinking Scale (OCDS). Cue induced OCDS will be measured after alcohol cues viewing. French version of OCDS is a self-administrated 14-items instrument assessing obsessive and compulsive characteristics of drinking-related thoughts, urge to drink or craving, and ability to resist those thoughts and urges. This scale is scored out of 56, higher scores are considered worse. Alcohol cues consisted of a selection of 60 alcohol-related pictures (beverage, drinking-related behaviors, alcohol-related cues) from the Geneva Appetitive alcohol Pictures . The same diaporama will be used for all visits in all centers.
Alcohol cue induced craving using the Cue induced Obsessive Compulsive Drinking Scale (OCDS) | at 1 month after the end of rTMS sessions
  Evaluated by Cue induced Obsessive Compulsive Drinking Scale (OCDS). Cue induced OCDS will be measured after alcohol cues viewing. French version of OCDS is a self-administrated 14-items instrument assessing obsessive and compulsive characteristics of drinking-related thoughts, urge to drink or craving, and ability to resist those thoughts and urges. This scale is scored out of 56, higher scores are considered worse. Alcohol cues consisted of a selection of 60 alcohol-related pictures (beverage, drinking-related behaviors, alcohol-related cues) from the Geneva Appetitive alcohol Pictures . The same diaporama will be used for all visits in all centers.
Alcohol cue induced craving using the Cue induced Obsessive Compulsive Drinking Scale (OCDS) | at 3 months after the end of rTMS sessions
  Evaluated by Cue induced Obsessive Compulsive Drinking Scale (OCDS). Cue induced OCDS will be measured after alcohol cues viewing. French version of OCDS is a self-administrated 14-items instrument assessing obsessive and compulsive characteristics of drinking-related thoughts, urge to drink or craving, and ability to resist those thoughts and urges. This scale is scored out of 56, higher scores are considered worse. Alcohol cues consisted of a selection of 60 alcohol-related pictures (beverage, drinking-related behaviors, alcohol-related cues) from the Geneva Appetitive alcohol Pictures . The same diaporama will be used for all visits in all centers.
Change in Alcohol cue induced craving using a Visual Analogic Scale (VAS) | From baseline to the last rTMS session after the end of rTMS sessions
  Change in cue induced craving Visual Analogic Scale (VAS) from baseline to the last rTMS session.
  Cue induced craving VAS will be measured after alcohol cues viewing at baseline and then daily on the morning just before rTMS sessions. The VAS is scored out of 10, higher scores are considered worse. Alcohol cues will be the same as for OCDS.
Alcohol cue induced craving using a Visual Analogic Scale (VAS) | At 1 month after the end of rTMS sessions
  The VAS is scored out of 10, higher scores are considered worse. Alcohol cues will be the same as for OCDS.
Alcohol due induced craving using a Visual Analogic Scale (VAS) | At 3 months after the end of rTMS sessions
  The VAS is scored out of 10, higher scores are considered worse. Alcohol cues will be the same as for OCDS.
Number of impaired measures on the Grefex batery (executive functions) | 1 month after the end of rTMS sessions
  Executive performance will be evaluated by the number of impaired measures on the Grefex battery : Stroop test, Wisconsin Test, Trail Making Test, verbal fluency, 6 elements, Brixton test and Dual task Baddeley test. Upon these 7 tests, 19 index will be measured (number of errors, time to make the task .). Each measure will be considered as impaired if it is below 1.65 SD. Number of impaired measures will be recorded for each patient.
Stroop test | 1 month after the end of rTMS sessions
  Stroop test will be performed 1 month after the end of the rTMS sessions. The stroop test assess the cognitive inhibition. Time and number of non-corrected errors will be reported for each conditions 1) denomination 2) reading 3) interference.
Trail making test | 1 month after the end of rTMS sessions
  Trail making test will be performed 1 month after the end of the rTMS sessions. The trail making test assess the mental flexibility. Time and number of errors will be reported for the trail making test A and the trail making test B. For this last condition, the number of perserverations will be also reported.
Verbal fluency | 1 month after the end of rTMS sessions
  Verbal fluency will be performed 1 month after the ned of the rTMS sessions. The verbal fluency assess the lexical generation ability. The number of words produced will be reported.
Wisconsin Test | 1 month after the end of rTMS sessions
  Wisconsin test will be performed 1 month after the ned of the rTMS sessions. The Wisconsin test assess the ability of deduction and rules maintenance. Number of correct categories, number of errors and number of perseverations will be reported.
Brixton test | 1 month after the end of rTMS sessions
  Brixton test test will be performed 1 month after the ned of the rTMS sessions. The Brixton test assess the deduction abilify of working rules. Number of errors will be reported.
6 elements | 1 month after the end of rTMS sessions
  6 elements test will be performed 1 month after the ned of the rTMS sessions. The 6 elements test assess the planning and organization ability of the behavior. Ranking score will be reported.
Dual task Baddeley test | 1 month after the end of rTMS sessions
  Dual task Baddeley testwill be performed 1 month after the end of the rTMS sessions. The Dual task Baddeley assess the working memory. Mu index will be reported.
Quality of life assessed by the Quality of life Scale (AQoLS) | At 1 month after the end of rTMS sessions
  Quality of life will be evaluated with Alcohol Quality of Life Scale (AQoLS) French version. This scale is a self-administrated 34-item questionnaire measuring health-related quality of life. The questionnaire explores 7 domains, i.e. activities, relationships, self-esteem, negative emotions, living conditions, control and sleep. The total score was obtained by summing all items, and the theoretical range was therefore 0-102; higher scores are considered better.
Quality of life assessed by the Quality of life Scale (AQoLS) | At 3 months after the end of rTMS sessions
  Quality of life will be evaluated with Alcohol Quality of Life Scale (AQoLS) French version. This scale is a self-administrated 34-item questionnaire measuring health-related quality of life. The questionnaire explores 7 domains, i.e. activities, relationships, self-esteem, negative emotions, living conditions, control and sleep. The total score was obtained by summing all items, and the theoretical range was therefore 0-102; higher scores are considered better.
% rTMS stimulation performed with optimal stimulation parameters | At the end of rTMS treatment
  Achievement of optimal stimulation parameters will be assessed for each patient by the percentage of sessions performed with the theoretical threshold (110%).
Percentage of rTMS sessions performed. | At the end of rTMS treatment
  Treatment compliance will be assessed by the percentage of rTMS sessions performed.
Percentage of participants experiencing sides effect | 3 months at the end of rTMS treatment
  rTMS security will be assessed by the percentage of patients experiencing sides effects during the study and their nature: seizure induction, transient acute hypomania induction, syncope, transient headache, local pain, neck pain, toothache, paresthesia, transient hearing changes, other.

CONTACTS AND LOCATIONS:
Overall Officials: Fanny LEVY, Docteur, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Universitaire Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request. The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal